CLINICAL TRIAL: NCT03735758
Title: Quality of Life in Patients With Non-adipocyte Soft Tissue Sarcoma Under Palliative Chemotherapy or Pazopanib - a Randomized, Controlled Trial
Brief Title: Quality of Life in Patients With Non-adipocyte Soft Tissue Sarcoma Under Palliative Chemotherapy or Pazopanib
Acronym: PazoQoL
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: problems with recruiting
Sponsor: GWT-TUD GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PazoQoL
Record Dates: First submitted 2018-11-07; First posted 2018-11-08 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2019-09

CONDITIONS: Soft Tissue Sarcoma Adult
Keywords: in-label prescription; Quality of Life; pazopanib; chemotherapy
MeSH Terms: interventions — pazopanib

STUDY DESIGN:
Intervention Model Description: multicentric, controlled, randomized, open Label, parallel-group, prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pazopanib (Experimental): Pazopanib; 800 mg; daily; oral
  Interventions: Drug: pazopanib or guideline conform chemotherapy
- Chemotherapy (Active Comparator): Guideline-conform chemotherapy
  Interventions: Drug: pazopanib or guideline conform chemotherapy

INTERVENTIONS:
Drug: pazopanib or guideline conform chemotherapy — Pazopanib (800mg/each day) or guideline conform chemotherapy

SUMMARY:
Finding the balance between toxicity and benefit should be the major goal when negotiating about the therapeutic regimen. This becomes nowadays even more important, since there are emerging options in the field of sarcoma therapy. Especially in the palliative treatment of sarcoma patients, knowing that na single drug can provide an overall survival benefit, physicians have to incorporate the patient's preferences and goals in life when consulting them.

The study will allow patients with several types of soff tissue sarcoma to be included. After progression under current therapy, the patient will be randomized in a 1:1 fashion and allocated to either pazopanib or investigator's choice. Quality of life (QoL) and other secondary outcome measures will be recorded continuously. The aim of the study is to assess patient reported outcomes (PROs), which should be the primary aim when treating these patients.

DETAILED DESCRIPTION:
Primary objectives

• Assess the overall quality of life (QoL) under treatment with pazopanib or physician-preferred chemotherapy after 9 weeks

Secondary objectives

* Assess the overall QoL under treatment with pazopanib compared with the physician's preference of chemotherapy three times in Cycle 1 and Cycle 3
* intergroup evaluation of pain

  * intergroup evaluation of fatigue and its different categories (physical, mental, cognitive, emotional)
  * intergroup evaluation of anorexia/cachexia
  * intergroup evaluation of satisfaction with care
  * Evaluation of the association of QoL with criteria of response
  * Evaluation of the QoL of all patients during follow up (FU) intergroup evaluation of treatment effects on survival
* Evaluation of the prediction of severe early toxicity in elderly patients receiving palliative therapy
* Safety and efficacy of the different treatment regimens

Exploratory Endpoints:

* QLQ-C30 sum score AUC (Area Under the Curve)
* Questionnaire Completion Times of QLQ-C30
* Questionnaire Completion of Time Tradeoff

ELIGIBILITY:
Inclusion Criteria:

* The informed consent form must be signed before any study specific tests or procedures are done
* Male or female patients aged 18 years and older at the first screening visit
* Histologically confirmed diagnosis of advanced or metastatic non adipocyte soft tissue sarcoma (STS)
* Suitable for treatment with pazopanib in an in-label prescription
* Patients with a life expectancy of at least 6 months
* Eastern Co-operative Oncology Group (ECOG) performance status 0-2
* Adequate organ function as given in Table 1
* For patients with previous anthracycline therapy a normal heart function needs to be documented with an left ventricular ejection fraction (LVEF) of minimal 50% (echocardiogram)
* Patients must be willing and able to fill in the Quality of live (QoL) questionnaires using a tablet PC
* Ability to understand and follow study-related instructions
* Confirmation of the subject's health insurance coverage prior to the first visit

Exclusion Criteria:

* Pretreatment with pazopanib
* Contraindications according to the local Summary of product characteristics ( SmPC) of Votrient®
* Patients having to following STS specific tumors

  * adipocyte sarcoma including all subtypes,
  * all rhabdomyosarcoma, which are not alveolar or pleomorph
  * Chondrosarcoma
  * Osteosarcoma
  * Ewing-tumors, i.e. primitive neuroectodermal tumors (PNET), gastrointestinal stromal tumor (GIST)
  * Dermatofibrosarcoma protuberans
  * inflammatory myofibroblastic sarcoma
  * Malignant mesothelioma
  * Mixed mesenchymal and epidermal tumors of the uterus Other malignant underlying diseases with the exception of the following:
  * Free of disease for at least 3 years
  * Completely resected, non-melanoma skin cancer
  * Successfully treated carcinoma in situ
  * Patients with metastases of the central nervous system (CNS) at screening, which are asymptomatic AND do not require treatment with steroids or enzyme-inducing anticonvulsant drugs
  * Patients with metastases of the CNS, which are already treated (operation and/or radiotherapy, radiosurgery or gamma-knife)
* Major surgery or trauma within 28 days before the first dose of study medication and / or presence of a non-healing wound, fracture, or ulcer
* Clinical indications of an active bleeding or a bleeding diathesis
* Known endobronchial lesions or lesions that infiltrate the large pulmonary artery
* Hemoptysis of> 2.5 mL within 8 weeks before the first dose of study drug
* Existing uncontrolled infection
* Heart rate-corrected QT-time according to the Fridericia's-formula (QTcF) 450 ms in males and 460 ms in females
* History of one or more of the following cardiovascular diseases within the last 6 months:

  * Cardiac angioplasty or coronary stent
  * Myocardial infarction
  * Unstable angina pectoris
  * Coronary artery bypass surgery
  * Symptomatic peripheral arterial disease
* Cardiac insufficiency New York Heart Association (NYHA) functional dass III or IV
* Poorly controlled hypertension defined as systolic blood pressure 140 mmHg or diastolic blood pressure 90 mmHg
* History of cerebrovascular disease, including transient ischemic attacks (TIA), pulmonary embolism or untreated deep vein thrombosis within 6 months prior to study entry. Patients with deep vein thrombosis who have received therapeutic anticoagulation for a minimum of 6 weeks might be included in the study.
* Clinically significant gastrointestinal changes that increase the risk of gastrointestinal bleeding
* Clinically significant gastrointestinal changes that may affect the absorption of the study drugs
* Treatment with any of the following anti-neoplastic therapies:

  * Irradiation or Tumor embolization within 14 days prior to the first dose of study drug
  * Chemotherapy, immunotherapy, biological therapy, study medication or hormonal therapy within 14 days or 5 half lives of substance (whichever is langer) prior to the first dose of study drug
* If the discontinuation of prohibited medication (see Section 6.9) at least 14 days or 5 half-lives of substance (whichever is langer) prior to the first dose of pazopanib is medically not acceptable or refused by the patient
* A history of hypersensitivity to any of the study drugs or their ingredients or to drugs with similar chemical structure
* Addiction or other diseases that preclude the patient from appropriately assessing the nature and scope as well as possible consequences of the clinical trial
* Pregnant or breast-feeding women
* Women of childbearing potential unless women who meet the following criteria:

  * Post-menopausal (12 months natural amenorrhea without any application of a hormonal contraceptive or hormonal substitution therapy))
  * Postoperatively (6 weeks after bilateral ovariectomy with or without hysterectomy)
  * Regular and correct use of a contraceptive method with error rate <1% per year such as implants, depot injections, oral contraceptives or intrauterine devices during treatment and up 6 months after end of treatment
  * Sexual abstinence
  * Vasectomy of the partner
* Men of sexual activity with women of childbearing potential who are not willing to use an effective barrier method of contraception during and up to 6 months after the end of therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2020-10-06 (Actual)

PRIMARY OUTCOMES:
The sum scores of the overall Quality of live (Qol) recorded with the questionaire "QLQ-C30" in patients with pazopanib versus chemotherapy treatment. | 9 weeks
  The 30 items of the QLQ-C30 questionaire distribute in diverse subscales (for example: cognitive function, pain and emotional function). The sum score of QLQ-C30 is generated by average of the normative values of all subscales. The higher the sum score the higher the Quality of live (Qol).

CONTACTS AND LOCATIONS:
Overall Officials: Markus Schuler, Dr., Principal Investigator — Helios Klinikum Emil von Behring
Locations (10):
- Germany (10):
  - Sarkomzentrum Berlin-Brandenburg, Bad Saarow
  - Charite, Berlin
  - Vivantes Klinikum Spandau, Berlin
  - Universitätsklinikum Dresden, Dresden
  - Uniklinik Frankfurt, Frankfurt
  - Medizinische Hochschule Hannover, Hanover
  - Uniklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Mannheim, Mannheim
  - Uniklinik Großhadern, München
  - Universitätsklinik der Paracelsus Privatuniversität Nürnberg, Nuremberg